CLINICAL TRIAL: NCT02951910
Title: A Study of the Effect of Zinc-Hyaluronate on Ocular Surface Sensations in Patients With Dry Eye
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Kovács Illés, Assistant professor of Ophthalmology, Semmelweis University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SemmelweisU
Record Dates: First submitted 2016-10-28; First posted 2016-11-01 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Patients receiving zinc-hyaluronate eye drop
  Interventions: Device: Ophylosa tear supplement

INTERVENTIONS:
Device: Ophylosa tear supplement — Tear film dynamics is assessed by non-invasive tear film breakup time (NI-BUT) in parallel with continuous recordings of ocular sensations during forced blinking. Corneal sensitivity thresholds to selective stimulation of corneal mechanonociceptors, thermal receptors and chemical nociceptors are assessed using the Belmonte gas esthesiometer. All baseline measurements are repeated after one month of tear supplementation with zinc-hyaluronate (Ophylosa eye drop) 4x/day

SUMMARY:
Hyaluronic acid, a natural polymer, helps to maintain ocular surface hydration and can already be found in several artificial tears recommended to alleviate symptoms of dry eye. A recent hyaluronate modification involves zinc-hyaluronate complex formation by adding zinc-chloride to an aqueous sodium-hyaluronate resulting in a very stable molecular structure, which functions as both a mechanical barrier and a biocompatible film on the ocular surface. Apart from its beneficial elastoviscous characteristics, previous results indicate that hyaluronate can also reduce the excitability of the peripheral nociceptor endings underlying pain. Although hyaluronate is widely used in artificial tears to improve tear film stability, its effect on ocular surface sensitivity was not evaluated in patients with dry eye. The aim of this study is to investigate the characteristics of ocular surface sensations and corneal sensitivity in dry eye patients before and after long-term tear supplementation with zinc-hyaluronate.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had been diagnosed as having dry eye symptoms for at least 3 months, with an OSDI score of ≥13 evaluated by the questionnaire of Ocular Surface Disease Index (OSDI)

Exclusion Criteria:

* Subjects with ophthalmic conditions other than dry eye or systemic disease including blepharitis, meibomitis, lid abnormalities as well as contact lens wearers

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-07; Primary Completion 2016-08 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change in OSDI (Ocular Surface Disease Index) score | 1 month
  The change in OSDI (Ocular Surface Disease Index) score will be assessed using the specific OSDI questionnaire

SECONDARY OUTCOMES:
Change in corneal sensitivity to selective stimulation | 1 month
  Corneal sensitivity to selective (thermal, mechanical, chemical) stimulation will be assessed using the noncontact Belmonte gas esthesiometer. Mechanical, chemical (CO2 in air), and cold stimuli were used during three-second air pulses of adjustable flow rate, composition (CO2%) and temperature.The good reproducibility of mechanical, heat and chemical threshold measurements using noncontact esthesiometers has been previously reported in several studies.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perenyi K, Dienes L, Kornafeld A, Kovacs B, Kiss HJ, Szepessy Z, Nagy ZZ, Barsi A, Acosta MC, Gallar J, Kovacs I. The Effect of Tear Supplementation with 0.15% Preservative-Free Zinc-Hyaluronate on Ocular Surface Sensations in Patients with Dry Eye. J Ocul Pharmacol Ther. 2017 Jul/Aug;33(6):487-492. doi: 10.1089/jop.2016.0194. Epub 2017 Apr 4. PMID 28375789